CLINICAL TRIAL: NCT01530347
Title: Assessing Feasibility of Non-invasive Breath Based Acetone Meter -Easy Check- Relative to Finger Capillary Blood Glucose and Beta Hydroxybutyrate Reference
Brief Title: Non Invasive Breath Based Acetone-meter- Easy Check
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Per sponsor decision to stop the development of the study device
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: rmc006631ctil
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Type 1 Diabetes
Keywords: Glucose monitoring; non-invasive glucometer; Self glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Easy Check versus reference glucometer and blood ketone meter (Experimental): Collection of paired measurements of capillary blood glucose using reference method (approved glucometer)and blood beta Hydroxybutyrate (approved ketone meter) and data generated by the non invasive study device
  Interventions: Device: Easy Check

INTERVENTIONS:
Device: Easy Check — Collection of paired measurements of capillary blood glucose using reference method and data generated by the non invasive study device. Samples will be obtained at specific time points during 4 hours: at fasting, and after consuming standard liquid meal at 60, 120, 180 and 240 minutes.

SUMMARY:
Segment 1- this segment will include two main steps:

Step 1-Calibration: During this step we plan to collect paired measurements of capillary blood glucose using reference method and data generated by the non invasive study device. Samples will be obtained at specific time points during 4 hours: at fasting, and after consuming standard liquid meal at 60, 120, 180 and 240 minutes. At each time point capillary blood glucose will be measured using the invasive reference method. The paired reference and study device data will be analyzed using multivariate regression model to formulate a calibration algorithm model. This model will convert the acetone values measured by study device to blood glucose values.

step 2-Validation: During this segment the second step of this segment we plan to evaluate the validity and reliability of the non-invasive breath-based glucometer compared to standard invasive reference glucometer. Results will be compared using a Clark error grid.

Segment 2- During this segment we plan to collect paired measurements of capillary blood glucose beta Hydroxybutyrate using reference method and acetone values generated by the non invasive breath based study device. Samples will be obtained at specific time points during 4 hours after overnight fasting, while basal insulin will be suspended, which is accepted to produce ketosis.

ELIGIBILITY:
Inclusion Criteria:

* Signing an inform consent form
* Type 1 diabetes diagnosed at least 12 months prior to study inclusion
* Males aged > 18 years old
* 23< BMI < 28 (segment 1 only)
* Treatment with insulin pump (segment 2 only)
* Willing to perform all study related procedures

Exclusion Criteria:

* Psychiatric disorder
* Patients with one or more of the following diseases: malignancy, myocardial insufficiency, nephrologic disease or any other chronic disease
* Patients who are not willing or are not capable of performing the protocol requirements
* Participating in another study that includes investigational drug or investigational equipment
* Patients who are under low carbohydrate diet
* Patients who are known as heavy alcohol drinkers

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
correlation between the acetone values generated by study device and blood beta Hydroxybutyrate | up to 30 weeks
correlation between the acetone values generated by study device and blood glucose | up to 30 weeks
correlation between the acetone values generated by study device and HbA1c | up to 30 weeks
correlation between the acetone values generated by study device and oxygen | up to 30 weeks

SECONDARY OUTCOMES:
Clarke Error Grid (segment 1 only) | up to 30 weeks
  The Clarke Error Gride breaks down a scatter plot of a reference glucose meter and an evaluated glucose meter into five regions:
  values within 20% of the reference meter, values outside of 20% but would not lead to inappropriate treatment,points leading to unnecessary treatment,points indicating a potentially dangerous failure to detect hypoglycemia or hyperglycemia and points that would confuse treatment of hypoglycemia for hyperglycemia and vice-versa.

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, Principal Investigator — Rabin Medical Center
Locations (1):
- Schneider Children's Medical Center, Petah Tikva, Israel